CLINICAL TRIAL: NCT00031200
Title: MRI Derived Organ & Tissue Mass Changes With Weight Loss - Ancillary to Look AHEAD
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 991; R01HL070298 (NIH)
Record Dates: First submitted 2002-02-27; First posted 2002-02-28 (Estimated); Last update posted 2016-07-29 (Estimated); Status verified 2008-01

CONDITIONS: Cardiovascular Diseases; Atherosclerosis; Obesity; Diabetes Mellitus, Non-insulin Dependent; Heart Diseases; Myocardial Infarction; Diabetes Mellitus
MeSH Terms: conditions — Cardiovascular Diseases; Atherosclerosis; Obesity; Diabetes Mellitus, Type 2; Heart Diseases; Myocardial Infarction; Diabetes Mellitus

SUMMARY:
To investigate the composition and nature of weight loss and weight maintenance during the Look AHEAD trial. Also, to model changes in resting energy expenditure and changes in cardiac structure and function associated with weight loss.

DETAILED DESCRIPTION:
BACKGROUND:

Advances in science are often achieved with the development of technology that allows scientists to differentiate and refine concepts which were previously undifferentiated. The field of obesity research has progressed from simple measurement of weight loss to multi-compartment models of fat, fat-free mass and regional distribution of fat. An opportunity for further refinement now presents itself in that magnetic resonance imaging technology can be used to image individual organs and tissues. This presents the opportunity to investigate important unresolved questions. For example, information is lacking on the effects of weight loss on individual organs and tissues. The loss of fat free mass (FFM) cannot fully explain the reported decrease in resting energy expenditure (REE) that accompanies weight loss. Since the FFM compartment consists of numerous tissues and organs, each with a different oxidative metabolic capacity, the possibility exists that individual vital organs may change disproportionately to the change in total FFM with weight loss, thereby explaining reductions in REE post weight loss. Complete organ-tissue volume and mass reconstruction of most major compartments is now possible, using magnetic resonance imaging (MRI).

The study is ancillary to the Look AHEAD clinical trial which is sponsored primarily by the National Institute of Diabetes and Digestive and Kidney Diseases and secondarily by the National Heart, Lung, and Blood Institute, the National Institute of Nursing Research, the Office of Research on Women's Health, the National Center on Minority Health and Health Disparities, and the Centers for Disease Control and Prevention. The Look AHEAD study is a multicenter, randomized clinical trial to examine the long-term effects of a lifestyle intervention designed to achieve and maintain weight loss in overweight diabetics.

DESIGN NARRATIVE:

The study will describe the composition of weight loss in diabetic subjects at the tissue/organ level of body composition; specifically, to determine whether and to what degree different tissues and organs are conserved or lost in comparison to total fat free mass (FFM) change during weight loss. The study will also assess the effects of aging on organ and tissue mass in 50+ year old diabetic men and women in a control group. The study will test whether a portion of weight loss related changes in resting energy expenditure (REE) can be explained by changes in the relative fractions of body mass as high (brain, heart, liver, kidney) and low (skeletal muscle, adipose tissue) metabolic activity tissues with respect to oxidative metabolism in 50 plus year old diabetic men and women. A secondary aim is to assess the effects of weight loss on cardiac structure and function using cardiac gated MRI. Consenting, eligible Look AHEAD participants at St. Luke's and at the University of Pittsburgh will participate in MRI and REE tests. Seventy men and women will be measured, equally distributed between the two sites, and equally distributed between Lifestyle Intervention group and a Community Care group. Measures will be acquired at baseline, following one year of intervention (Year 1), and following one year of maintenance (Year 2), to produce a 2 X 3 factorial design.

ELIGIBILITY:
An estimated 140 obese, diabetic men and women, ages 45 or older. There will be 70 women (50%) and 20% minorities

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2001-09; Primary Completion 2007-02 (Actual); Study Completion 2007-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dympna Gallagher — St. Luke's-Roosevelt Hospital Center

REFERENCES:
- [Background] Gallagher D, Song MY. Evaluation of body composition: practical guidelines. Prim Care. 2003 Jun;30(2):249-65. doi: 10.1016/s0095-4543(03)00030-7. PMID 14567146
- [Background] He Q, Horlick M, Thornton J, Wang J, Pierson RN Jr, Heshka S, Gallagher D. Sex-specific fat distribution is not linear across pubertal groups in a multiethnic study. Obes Res. 2004 Apr;12(4):725-33. doi: 10.1038/oby.2004.85. PMID 15090643